CLINICAL TRIAL: NCT02971397
Title: Cytarabine Plus Continuous Infusion Daunorubicin Induction Therapy for Adults With Acute Myeloid Leukemia: A Feasibility Study With Cardiac MRI Monitoring
Brief Title: Cytarabine and Daunorubicin Hydrochloride in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00040792; NCI-2016-01464 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 22616 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-10-04; First posted 2016-11-23 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Biopsy; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cytarabine, daunorubicin hydrochloride, biopsy) (Experimental): INDUCTION: Patients receive cytarabine IV continuously over 24 hours on days 1-7 and daunorubicin hydrochloride IV continuously over 24 hours on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients then undergo bone marrow aspirate and biopsy on day 14. Patients with bone marrow cellularity >= 10% and > 5% leukemic blasts, may receive a second induction of cytarabine IV continuously over 24 hours on days 1-5 and daunorubicin hydrochloride IV continuously over 24 hours on days 1-2 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients achieving remission receive cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients with CBF AML may receive 4 courses of therapy.
  Interventions: Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies the side effects of cytarabine and daunorubicin hydrochloride and to see how well they work in treating patients with newly diagnosed acute myeloid leukemia. Drugs used in chemotherapy, such as cytarabine and daunorubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading, and may be safer for the heart.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety (at 3 months) and feasibility of administering daunorubicin hydrochloride (daunorubicin) as continuous infusion under the proposed treatment regimen.

SECONDARY OBJECTIVES:

I. To assess the safety (at 6 months) of administering daunorubicin as continuous infusion under the proposed treatment regimen.

II. To assess treatment outcomes (including complete remission [CR] and complete remission with incomplete recovery [CRi]) in patients with acute myeloid leukemia (AML) under the proposed treatment regimen.

III. To compare the concordance between magnetic resonance imaging (MRI) and echocardiogram (ECHO) in identifying cardiac toxicity, ie a reduction in left ventricular ejection fraction (LVEF) of >= 10% and ejection fraction (EF) =< 50% compared to baseline LVEF.

OUTLINE:

INDUCTION: Patients receive cytarabine intravenously (IV) continuously over 24 hours on days 1-7 and daunorubicin hydrochloride IV continuously over 24 hours on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients then undergo bone marrow aspirate and biopsy on day 14. Patients with bone marrow cellularity >= 10% and > 5% leukemic blasts, may receive a second induction of cytarabine IV continuously over 24 hours on days 1-5 and daunorubicin hydrochloride IV continuously over 24 hours on days 1-2 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients achieving remission receive cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients with core-binding factor (CBF) AML may receive 4 courses of therapy.

After completion of study treatment, patients are followed up for a minimum of 30 days, at 3 and 6 months, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have morphologically confirmed newly diagnosed acute myelogenous leukemia (AML) with blood or bone marrow disease; patients with only extramedullary disease in the absence of bone marrow or blood involvement are eligible; note: this protocol uses World Health Organization (WHO) diagnostic criteria for AML; patients with acute promyelocytic leukemia (APL, French-American-British Classification [FAB], M3) or blastic transformation of chronic myelogenous leukemia (CML) are not eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Patients with ECHO EF >= 45% within 28 days prior to registration
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Patients who have received prior induction chemotherapy for AML or myelodysplastic syndrome (MDS); temporary prior measures such as apheresis or hydroxyurea are allowed; patients who have received a limited and short-term exposure of ATRA (all trans retinoic acid) while AML-M3 (acute promyelocytic leukemia) was being ruled out, and which has been discontinued, will be eligible
* Patients receiving any other investigational agents
* Patients with prolonged corrected QT (QTc) interval (> 500 msec) determined by electrocardiogram (EKG) within 28 days prior to registration
* Patients not suitable for cardiac MRI; contraindications include:

  * Intracranial metal, pacemakers, defibrillators, functioning neurostimulator devices, or other implanted electronic devices
  * Ferromagnetic cerebral aneurysm clips, or other intraorbital/intracranial metal
  * Allergy to gadolinium or other severe drug allergies
  * Claustrophobia
  * Congestive heart failure (New York Heart Association [NYHA] class III or IV)
  * Significant valvular disease, or significant pulmonary disease requiring supplemental oxygen therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to daunorubicin or cytarabine
* Patients with documented central nervous system (CNS) involvement
* Patients who are known to be human immunodeficiency virus (HIV) positive (+) may be eligible providing they meet all of the following additional criteria within 28 days prior to registration:

  * CD4 cells >= 500/mm^3
  * Viral load of < 50 copies HIV messenger ribonucleic acid (mRNA)/mm^3 if on combination antiretroviral therapy (cART) or < 25,000 copies HIV mRNA if not on cART
  * No zidovudine or stavudine as part of cART Patients who are HIV+ and do not meet all of these criteria are not eligible for this study
* Patients with other uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued prior to beginning treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Change in incidence of cardiac toxicity, defined as reduction in LVEF of >= 10% compared to baseline LVEF and EF =< 50% on the follow-up scan, assessed using MRI | Baseline up to 3 months after last dose of study drug
  In addition to point estimates of these rates, 95% confidence intervals will be calculated.
Incidence of other unexpected toxicities, measured by Common Terminology Criteria for Adverse Events version 4.0 | Up to 6 months after last dose of study drug
  In addition to point estimates of these rates, 95% confidence intervals will be calculated.
Proportion of patients who complete the infusion therapy | Up to 4 months
  Will report these proportions with 95% confidence intervals.
Proportion of patients with study-related deviations | Up to 2 years
  Will report these proportions with 95% confidence intervals.
Change in incidence of cardiac toxicity, defined as reduction in LVEF of >= 10% compared to baseline LVEF and EF =< 50% on the follow-up scan, assessed using ECHO | Baseline up to 3 months after last dose of study drug
  In addition to point estimates of these rates, 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
Change in EF, assessed by MRI and ECHO | Baseline up to 6 months after last dose of study drug
  Will determine the correlation between ECHO and MRI assessments performed pre-chemotherapy. Will assess correlations between post-chemotherapy ECHO and MRI assessments. Will assess correlations between each of the time points. Paired t-tests will be performed to compare the actual values of each ECHO/MRI measurement to each other at each time point. Bland-Altman plots will be generated at baseline, follow-up and using the change in measure for each of the MRI/ECHO derived measures.
Change in incidence of cardiac toxicity, defined as reduction in LVEF of >= 10% compared to baseline LVEF and EF =< 50% on the follow-up scan, assessed using MRI and ECHO | Baseline up to 6 months after last dose of study drug
  Will determine the correlation between ECHO and MRI assessments performed pre-chemotherapy. Will assess correlations between post-chemotherapy ECHO and MRI assessments. Will assess correlations between each of the time points. Paired t-tests will be performed to compare the actual values of each ECHO/MRI measurement to each other at each time point. Bland-Altman plots will be generated at baseline, follow-up and using the change in measure for each of the MRI/ECHO derived measures.
Change in left ventricular end diastolic volume, assessed by MRI and ECHO | Baseline up to 6 months after last dose of study drug
  Will determine the correlation between ECHO and MRI assessments performed pre-chemotherapy. Will assess correlations between post-chemotherapy ECHO and MRI assessments. Will assess correlations between each of the time points. Paired t-tests will be performed to compare the actual values of each ECHO/MRI measurement to each other at each time point. Bland-Altman plots will be generated at baseline, follow-up and using the change in measure for each of the MRI/ECHO derived measures.
Change in left ventricular end systolic volume, assessed by MRI and ECHO | Baseline up to 6 months after last dose of study drug
  Will determine the correlation between ECHO and MRI assessments performed pre-chemotherapy. Will assess correlations between post-chemotherapy ECHO and MRI assessments. Will assess correlations between each of the time points. Paired t-tests will be performed to compare the actual values of each ECHO/MRI measurement to each other at each time point. Bland-Altman plots will be generated at baseline, follow-up and using the change in measure for each of the MRI/ECHO derived measures.
Change in myocardial strain, assessed by MRI and ECHO | Baseline up to 6 months after last dose of study drug
  Will determine the correlation between ECHO and MRI assessments performed pre-chemotherapy. Will assess correlations between post-chemotherapy ECHO and MRI assessments. Will assess correlations between each of the time points. Paired t-tests will be performed to compare the actual values of each ECHO/MRI measurement to each other at each time point. Bland-Altman plots will be generated at baseline, follow-up and using the change in measure for each of the MRI/ECHO derived measures.
Disease-free survival for those patients who achieve remission | From the date of CR until relapse from CR or death, assessed for up to 2 years
Induction death rate | Up to 28 days
Overall response rate, defined as CR + CRi | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayard Powell, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT02971397/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT02971397/ICF_001.pdf